CLINICAL TRIAL: NCT02291315
Title: Calcium Bioavailability of Cassia Leaves in Post-Menopausal Women
Brief Title: Calcium Absorption in Postmenopausal Thai Women
Status: Completed | Type: Observational
Sponsor: Cornell University (Other)
Collaborators: Ramathibodi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB #: MU 2007-145
Record Dates: First submitted 2014-11-10; First posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Fractional Calcium Absorption
Keywords: Triple Stable Isotope

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Test meal ingestion: On the morning of the absorption study, fasted women received 2 mg of 42Ca intravenously (in 5 ml of isotonic saline) over 5 minutes before being randomly assigned to receive either the milk or cassia meal first for breakfast and the milk or cassia meal second for lunch. The milk meal consisted of approximately 100 mg of fresh ultrahigh temperature (UHT) milk to which 2 mg of 44Ca was added and allowed to equilibrate for 12 h prior to ingestion and the cassia meal consisted of 142 g of cooked cassia to which 1 mg of 43Ca was extrinsically added.

SUMMARY:
Adequate calcium absorption is essential for reducing one's risk of developing osteoporosis. However, postmenopausal Thai women consume diets which are habitually low in calcium due to lactose intolerance and dietary patterns which typically do not include milk-based products. The primary goal of this study is to measure the fractional calcium absorption from milk and a commonly ingested green leafy vegetable (cassia) in postmenopausal Thai women with habitually low calcium intakes. The secondary objective is to determine associations between calcium absorption and biomarkers which impact vitamin D status and bone metabolism.

DETAILED DESCRIPTION:
Postmenopausal Thai women (n=22) will be recruited from the community surrounding Bangkok and Nakhon Pathon, Thailand. They will be invited to participate in an isotope study comparing the fractional calcium absorption from milk and cassia. Upon arrival, a fasting blood sample will be drawn on the morning of the absorption study to analyze serum markers of vitamin D and bone metabolism (25-hydroxy vitamin D [25OHD], parathyroid hormone [PTH], and beta-crossLaps) and to determine their impact on calcium absorption. Following this blood draw, women will receive a stable calcium isotope (42Ca) intravenously. Then for breakfast and lunch respectively, the women will be randomly assigned to orally ingest a stable calcium isotope from either the milk (44Ca) or cassia (43Ca) test meals. On day two, women will receive a breakfast, snack, and lunch meal. Urine samples will be collected over the entire 28 hour period and the 24-hr urine collection will be used to measure urinary calcium concentration and to calculate fractional calcium absorption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* At least 3 years postmenopausal

Exclusion Criteria:

* Diagnosed gastrointestinal or metabolic diseases known to interfere with calcium absorption and metabolism
* Women taking medications (including thiazide diuretics, hormonal replacement therapy, etc.) within two months prior to the study
* Women taking dietary supplements within two months prior to the study

Ages: 53 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Post-menopausal Thai women
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2007-07; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Fractional calcium absorption | 24 hours after the ingestion of the second test meal
  Urine samples will be collected over s 28 hour period post-dosing with collection ending 24 hours after the ingestion of the second test meal.

SECONDARY OUTCOMES:
The concentration of 25-hydroxy vitamin D (25OHD) in serum | Upon entry to the study, a 10 mL blood sample will be collected in a less than 2 hour time period.
  A fasting 10 mL blood sample will be collected upon entry into the study and used for determining the concentration of 25OHD in serum.
The concentration of parathyroid hormone (PTH) in serum | Upon entry to the study, a 10 mL blood sample will be collected in a less than 2 hour time period.
  A fasting 10 mL blood sample will be collected upon entry into the study and used for determining the concentration of PTH in serum.
The concentration of beta-crossLaps in serum | Upon entry to the study, a 10 mL blood sample will be collected in a less than 2 hour time period.
  A fasting 10 mL blood sample will be collected upon entry into the study and used for determining the concentration of beta-crossLaps in serum.

CONTACTS AND LOCATIONS:
Overall Officials: Prapaisri P. Sirichakwal, PhD, Principal Investigator — Mahidol University
Locations (1):
- Human Metabolic Research Unit, Ithaca, New York, United States

REFERENCES:
- [Derived] Sirichakwal PP, Kamchansuppasin A, Akoh CC, Kriengsinyos W, Charoenkiatkul S, O'Brien KO. Vitamin D Status Is Positively Associated with Calcium Absorption among Postmenopausal Thai Women with Low Calcium Intakes. J Nutr. 2015 May;145(5):990-5. doi: 10.3945/jn.114.207290. Epub 2015 Mar 25. PMID 25809682